CLINICAL TRIAL: NCT04221724
Title: A Multicomponent Physical Exercise Program: a Tool to Maintain Autonomy, Reduce Frailty and Improve Functionality in Nursing Homes. Interventional Single Group Study
Brief Title: Effects of Function-focused Multicomponent Physical Exercise Program. Interventional Single Group Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Itxaso Mugica Errazquin, Principal investigator, University of the Basque Country (UPV/EHU)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Functional-Ageing On
Record Dates: First submitted 2020-01-03; First posted 2020-01-09 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Activities of Daily Living; Frailty; Older Adults; Long Term Care
Keywords: Exercise; Physical Activity; Aging
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: Multicenter single group interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Multicomponent physical exercise intervention
  Interventions: Other: Multicomponent physical exercise program

INTERVENTIONS:
Other: Multicomponent physical exercise program — The intervention consists of a combined multicomponent exercise program (EP) carried out for 6 months that includes strength, balance, flexibility and functional exercises aimed to improve functioning on daily life activities. The EP will be divided into two parts:
  The first 3 months the EP aims to restore the physical condition through the multicomponent exercise program. This program will comprise of upper and lower body strengthening exercises, using external weights for 2-3sets of 8-12repetitions at a progressive intensity of 30-50% of 1RM. In addition, static balance and flexibility exercise will be performed.
  From 3th to 6th months, the objective will be to improve autonomy through the functional EP. Strength exercises intensity will be increased to 60-70% of 1-RM, 2-3sets of 8-12repetitions. Attention tasks, temporal space dissociation and dynamic balance exercises will be added to increase the intensity in balance exercises. Flexibility and fine handle will be also performed

SUMMARY:
The purpose of this research study is to determine whether a physical exercise program in nursing homes will maintain autonomy in activities of daily living, decrease vulnerability and improve physical, psychological and cognitive condition. An individualized and progressive multi-component physical exercise program focused on function has been designed to achieve this objective.

Participant will engage in an exercise program for 6 months in their nursing homes, in two sessions per week of 45-60 minutes

DETAILED DESCRIPTION:
Primary aim:

The major aim is to ascertain whether multicomponent exercise program focused on function can maintain autonomy in older adults living in nursing homes.

Secondary aims:

* To ascertain the influence of the evaluated exercise program on frailty, physical, psycho-affective and cognitive conditions in older people living in nursing homes.
* Analyze if the influence that the exercise program has had on dependence, frailty, physical, psycho-affective and cognitive condition is maintained after 6 months since the end of the program
* Examine the influence that the exercise program has on different clinical outcomes: falls, hospitalizations, visits to emergency service, the level of dependence, etc.

Design: experimental, multi-center and single-group physical exercise intervention

Intervention:

Combined multicomponent physical exercise program that includes strength, balance and flexibility exercises and performed in long term care homes focused on functionality on activities of daily living.

The first 3 months the exercise program aims to restore the physical condition through the multicomponent exercise program. Feasibility and safety of the multicomponent exercise program were ascertained in a previous study (Arrieta et al., 2018; Rodriguez-Larrad et al., 2017). This program will comprise of upper and lower body strengthening exercises, using external weights for 2-3 sets of 8-12 repetitions at a progressive incremental intensity of 30-50% of 1Repetition Maximum (RM). In addition, static balance and flexibility exercise will be performed.

From 3th to 6th months, the objective will be to improve autonomy in daily live activities through the functional exercise program. Strength exercises will be maintained with external weights and the intensity will be increased to 60-70% of 1-RM, 2-3 sets of 8-12 repetitions. Attention tasks, temporal space dissociation and dynamic balance exercises will be added to increase the difficulty and intensity in balance exercises. Flexibility and fine handle will be also performed.

This intervention is individualized for each participant and is adjusted progressively during the 6 months. Weekly, two sessions of one hour are held and are supervised by physiotherapists or specialists in sports sciences trained specifically for the program. An interval of at least 48h between training sessions will be respected.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥70years
* Scored ≥50 on the Barthel index
* Scored ≥20 on Mini Examen Cognoscitive test (MEC-35), validated and adapted Spanish version of Mini Mental State Examination
* Be able to stand up from the chair and walk 10 meters with or without one person/technical assistance.

Exclusion Criteria:

* If the participants are clinically unstable under the clinical judgment of the medical professionals of the reference center,
* If the risk of adverse effects is greater than the benefit
* If the participants have severe cognitive or psychiatric disorders.

Ages: 70 Years to 115 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Barthel Index | Changes from baseline to 3rd 6th and 12th month
  Autonomy on daily living activities will be analyzed using the Barthel index. The Barthel index is a questionnaire with 10 items that evaluates the autonomy of the participant in the activities of daily life and it will be evaluated with the reference caregiver in nursing home. The Barthel index evaluates the following items: Feeding, Bathing, Dressing, Grooming, Bowels, Bladder, Toilette use, Transfer, Walking and Stairs. This items are scored as follows: 0 points if it is totally dependent, 5 points if needs some help and 10 points if the participant is totally autonomous
Short Physical Performance Battery | Changes from baseline to 3rd 6th and 12th month
  Short Physical Performance Battery (SPPB) evaluates balance, gait ability, and leg strength using a single tool. The score for each part is given in categorical modality (0-4). This set of tests serves to predict falls, weakness and mortality. The best score will be 12 points and total score less than 10 points indicates frailty and high risk of disability. 1 point of change in the total score has demonstrated to be of clinical relevance.
Handgrip strength | Changes from baseline to 3rd 6th and 12th month
  To asses upper limbs strength (kg) will be used bilateral handgrip strength test by squeezing a dynamometer with maximum isometric effort for 5 seconds. It is a strong predictor of disability, morbidity, and mortality as well as one of the components of Fried's frailty phenotype. Ranges are corrected by BMI
Timed Up and Go Test | Changes from baseline to 3rd 6th and 12th month
  Timed Up and Go (TUG) is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. The cut-off value for the TUG is 12 seconds The test score also correlates well with gait speed and the Barthel Index.

SECONDARY OUTCOMES:
Fried frailty index | Changes from baseline to 3rd 6th and 12th month
  Fried index uses 5 criteria to define frailty: weight loss, exhaustion, physical activity, walk time and grip strength. Fulfilling three of these criteria indicates clinical frailty.
Tilburg frailty indicator | Changes from baseline to 3rd 6th and 12th month
  Tilburg indicator evaluates frailty through a self-reported questionnaire that includes physical, psychological and social domains. The score range is from 0 points to 15 points. High scores indicates higher frailty
Rockwood frailty phenotype | Changes from baseline to 3rd 6th and 12th month
  9 phenotype ranging from very fit to terminally ill are evaluated in Rockwood frailty scale.
Anthropometry-Weight | Changes from baseline to 3rd 6th and 12th month
  Weight (kg)
Anthropometry-Height | Changes from baseline to 3rd 6th and 12th month
  Height (m)
Body Mass Index | Changes from baseline to 3rd 6th and 12th month
  Body Mass Index (BMI), weight and height will be combined to report BMI in kg/m^2)
Anthropometry-Circumferences | Changes from baseline to 3rd 6th and 12th month
  Neck circumference, mid arm circumference and calf circumference (cm)
The Goldberg Anxiety and Depression Scale | Changes from baseline to 6th and 12th month
  The Goldberg Anxiety and Depression Scale will be used to assess affective state of anxiety and depression that includes nine depression and nine anxiety items from the last month. The cut-off points are ≥4 for the anxiety scale, and ≥2 for the depression scale.
The Spanish Subjective Happiness scale | Changes from baseline to 6th and 12th month
  The Spanish Subjective Happiness scale test will be used to analyze the perceived happiness. It ranges from 0 to 28 points in four questions. Higher punctuation means higher happiness level.
Quality of Life-Alzheimer Disease | Changes from baseline to 6th and 12th month
  Quality of Life-Alzheimer Disease (QoL-AD) test. Self-rated quality of life for people with cognitive impairments. The QoL-AD is comprised of 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores, ability to do things for fun, money and life as a whole). Response options include 1(poor), 2(fair), 3(good) and 4 (excellent), for a total score of 13-52, with higher scores indicating better QoL.
Montreal Cognitive Assessment test (MOCA test) | Changes from baseline to 6th and 12th month
  The cognitive function will be assessed by MOCA test. Montreal Cognitive Assessment cover domains: attention and concentration, executive functions, memory and language skills, conceptual thinking, calculation and orientation. The MOCA is a validated test in Spanish. It ranges from 0 ( worse score ) to 30 (best score). A score less than 26 indicates suggest mild cognitive decline
Pain level | Changes from baseline to 6th and 12th month
  Using a score from 0 points (lowest) to 10 points (highest) the participant will be asked to say how much it hurts in different parts of the body such as shoulders, elbows, wrists, neck, back, hips, knees and ankles
Clinical outcomes-Number of falls | The data will be collected one year and 6 months before starting the project, at intervention baseline, at 6 months and at 12 months
  Number of falls will be assessed with a clinical questionnaire
Clinical outcomes-visits to the emergency service | The data will be collected one year and 6 months before starting the project, at intervention baseline, at 6 months and at 12 months
  Visits to the emergency service will be assessed with a clinical questionnaire
Clinical outcomes-hospital admissions | The data will be collected one year and 6 months before starting the project, at intervention baseline, at 6 months and at 12 months
  Hospital admissions will be assessed with a clinical questionnaire
Clinical outcomes-functional impairment | The data will be collected one year and 6 months before starting the project, at intervention baseline, at 6 months and at 12 months
  Functional impairment after hospitalization will be assessed with a clinical questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jon Irazusta Astiazaran, Professor, Study Director — University of the Basque Country (UPV/EHU); Ana Rodriguez Larrad, PhD, Study Director — University of the Basque Country (UPV/EHU)
Locations (1):
- Basque Country University, Leioa, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Larrad A, Arrieta H, Rezola C, Kortajarena M, Yanguas JJ, Iturburu M, Susana MG, Irazusta J. Effectiveness of a multicomponent exercise program in the attenuation of frailty in long-term nursing home residents: study protocol for a randomized clinical controlled trial. BMC Geriatr. 2017 Feb 23;17(1):60. doi: 10.1186/s12877-017-0453-0. PMID 28231827
- [Background] Rezola-Pardo C, Rodriguez-Larrad A, Gomez-Diaz J, Lozano-Real G, Mugica-Errazquin I, Patino MJ, Bidaurrazaga-Letona I, Irazusta J, Gil SM. Comparison Between Multicomponent Exercise and Walking Interventions in Long-Term Nursing Homes: A Randomized Controlled Trial. Gerontologist. 2020 Sep 15;60(7):1364-1373. doi: 10.1093/geront/gnz177. PMID 31845733
- [Background] Arrieta H, Rezola-Pardo C, Kortajarena M, Hervas G, Gil J, Yanguas JJ, Iturburu M, Gil SM, Irazusta J, Rodriguez-Larrad A. The impact of physical exercise on cognitive and affective functions and serum levels of brain-derived neurotrophic factor in nursing home residents: A randomized controlled trial. Maturitas. 2020 Jan;131:72-77. doi: 10.1016/j.maturitas.2019.10.014. Epub 2019 Nov 5. PMID 31787150
- [Background] Rezola-Pardo C, Arrieta H, Gil SM, Zarrazquin I, Yanguas JJ, Lopez MA, Irazusta J, Rodriguez-Larrad A. Comparison between multicomponent and simultaneous dual-task exercise interventions in long-term nursing home residents: the Ageing-ONDUAL-TASK randomized controlled study. Age Ageing. 2019 Nov 1;48(6):817-823. doi: 10.1093/ageing/afz105. PMID 31595289
- [Background] Arrieta H, Rezola-Pardo C, Gil SM, Virgala J, Iturburu M, Anton I, Gonzalez-Templado V, Irazusta J, Rodriguez-Larrad A. Effects of Multicomponent Exercise on Frailty in Long-Term Nursing Homes: A Randomized Controlled Trial. J Am Geriatr Soc. 2019 Jun;67(6):1145-1151. doi: 10.1111/jgs.15824. Epub 2019 Mar 19. PMID 30891748
- [Background] Rezola-Pardo C, Arrieta H, Gil SM, Yanguas JJ, Iturburu M, Irazusta J, Sanz B, Rodriguez-Larrad A. A randomized controlled trial protocol to test the efficacy of a dual-task multicomponent exercise program in the attenuation of frailty in long-term nursing home residents: Aging-ONDUAL-TASK study. BMC Geriatr. 2019 Jan 8;19(1):6. doi: 10.1186/s12877-018-1020-z. PMID 30626341
- [Background] Arrieta H, Rezola-Pardo C, Echeverria I, Iturburu M, Gil SM, Yanguas JJ, Irazusta J, Rodriguez-Larrad A. Physical activity and fitness are associated with verbal memory, quality of life and depression among nursing home residents: preliminary data of a randomized controlled trial. BMC Geriatr. 2018 Mar 27;18(1):80. doi: 10.1186/s12877-018-0770-y. PMID 29580209
- [Background] Arrieta H, Rezola-Pardo C, Gil SM, Irazusta J, Rodriguez-Larrad A. Physical training maintains or improves gait ability in long-term nursing home residents: A systematic review of randomized controlled trials. Maturitas. 2018 Mar;109:45-52. doi: 10.1016/j.maturitas.2017.12.003. Epub 2017 Dec 6. PMID 29452781
- [Background] Arrieta H, Rezola-Pardo C, Zarrazquin I, Echeverria I, Yanguas JJ, Iturburu M, Gil SM, Rodriguez-Larrad A, Irazusta J. A multicomponent exercise program improves physical function in long-term nursing home residents: A randomized controlled trial. Exp Gerontol. 2018 Mar;103:94-100. doi: 10.1016/j.exger.2018.01.008. Epub 2018 Jan 8. PMID 29326087
- [Background] de Souto Barreto P, Morley JE, Chodzko-Zajko W, H Pitkala K, Weening-Djiksterhuis E, Rodriguez-Manas L, Barbagallo M, Rosendahl E, Sinclair A, Landi F, Izquierdo M, Vellas B, Rolland Y; International Association of Gerontology and Geriatrics - Global Aging Research Network (IAGG-GARN) and the IAGG European Region Clinical Section. Recommendations on Physical Activity and Exercise for Older Adults Living in Long-Term Care Facilities: A Taskforce Report. J Am Med Dir Assoc. 2016 May 1;17(5):381-92. doi: 10.1016/j.jamda.2016.01.021. Epub 2016 Mar 21. PMID 27012368
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209
- [Background] Crocker T, Young J, Forster A, Brown L, Ozer S, Greenwood DC. The effect of physical rehabilitation on activities of daily living in older residents of long-term care facilities: systematic review with meta-analysis. Age Ageing. 2013 Nov;42(6):682-8. doi: 10.1093/ageing/aft133. Epub 2013 Sep 4. PMID 24004604
- [Background] Brett L, Traynor V, Stapley P. Effects of Physical Exercise on Health and Well-Being of Individuals Living With a Dementia in Nursing Homes: A Systematic Review. J Am Med Dir Assoc. 2016 Feb;17(2):104-16. doi: 10.1016/j.jamda.2015.08.016. Epub 2015 Oct 1. PMID 26432622
- [Background] Zucchella C, Bartolo M, Bernini S, Picascia M, Sinforiani E. Quality of life in Alzheimer disease: a comparison of patients' and caregivers' points of view. Alzheimer Dis Assoc Disord. 2015 Jan-Mar;29(1):50-4. doi: 10.1097/WAD.0000000000000050. PMID 24936799
- [Background] Kasper JD, Black BS, Shore AD, Rabins PV. Evaluation of the validity and reliability of the Alzheimer Disease-related Quality of Life Assessment Instrument. Alzheimer Dis Assoc Disord. 2009 Jul-Sep;23(3):275-84. doi: 10.1097/WAD.0b013e31819b02bc. PMID 19812471
- [Background] Maurer C, Draganescu S, Mayer H, Gattinger H. Attitudes and needs of residents in long-term care facilities regarding physical activity-A systematic review and synthesis of qualitative studies. J Clin Nurs. 2019 Jul;28(13-14):2386-2400. doi: 10.1111/jocn.14761. Epub 2019 Jan 15. PMID 30589972
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. Determinants of frailty. J Am Med Dir Assoc. 2010 Jun;11(5):356-64. doi: 10.1016/j.jamda.2009.11.008. PMID 20511103
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Extremera, N., & Fernández-Berrocal, P. (2014). The Subjective Happiness Scale: Translation and preliminary psychometric evaluation of a Spanish version. Social Indicators Research, 119(1), 473-481.
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Lazowski DA, Ecclestone NA, Myers AM, Paterson DH, Tudor-Locke C, Fitzgerald C, Jones G, Shima N, Cunningham DA. A randomized outcome evaluation of group exercise programs in long-term care institutions. J Gerontol A Biol Sci Med Sci. 1999 Dec;54(12):M621-8. doi: 10.1093/gerona/54.12.m621. PMID 10647968
- [Background] Toots A, Littbrand H, Lindelof N, Wiklund R, Holmberg H, Nordstrom P, Lundin-Olsson L, Gustafson Y, Rosendahl E. Effects of a High-Intensity Functional Exercise Program on Dependence in Activities of Daily Living and Balance in Older Adults with Dementia. J Am Geriatr Soc. 2016 Jan;64(1):55-64. doi: 10.1111/jgs.13880. PMID 26782852
- [Background] Rydwik E, Frandin K, Akner G. Effects of physical training on physical performance in institutionalised elderly patients (70+) with multiple diagnoses. Age Ageing. 2004 Jan;33(1):13-23. doi: 10.1093/ageing/afh001. PMID 14870716
- [Background] Cichocki M, Quehenberger V, Zeiler M, Adamcik T, Manousek M, Stamm T, Krajic K. Effectiveness of a low-threshold physical activity intervention in residential aged care--results of a randomized controlled trial. Clin Interv Aging. 2015 May 21;10:885-95. doi: 10.2147/CIA.S79360. eCollection 2015. PMID 26056438
- [Background] Jansen CP, Classen K, Wahl HW, Hauer K. Effects of interventions on physical activity in nursing home residents. Eur J Ageing. 2015 May 8;12(3):261-271. doi: 10.1007/s10433-015-0344-1. eCollection 2015 Sep. PMID 28804359
- [Derived] Mugica-Errazquin I, Irazusta J, Kortajarena M, Elosegi S, Wu B, Qi X, Rodriguez-Larrad A, Rezola-Pardo C. Maintaining daily living activities in older adults: The impact of a functional exercise program in long-term nursing homes. A single-group pre-post intervention. Geriatr Nurs. 2024 Nov-Dec;60:215-224. doi: 10.1016/j.gerinurse.2024.09.003. Epub 2024 Sep 14. PMID 39278126